CLINICAL TRIAL: NCT03467971
Title: A Randomized, Open-label, Single Dose, 2x2 Crossover Trial to Evaluate the Food Effect on the Bioavailability of a Metformin/Gliclazide Fixed Combination Tablet (1000 mg /30 mg MR) Given in Fasting and Fed Conditions to Healthy Volunteers
Brief Title: A Study to Assess the Food Effect on Bioavailability of Metformin/Gliclazide in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: EMR200763_004
Record Dates: First submitted 2018-03-12; First posted 2018-03-16 (Actual); Results first posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-04

CONDITIONS: Healthy
Keywords: Metformin; Bioavailability; Food effect; Pharmacokinetics
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Metformin-Gliclazide (fasted), Then Metformin-Gliclazide (fed) (Experimental): Participants received single dose of Metformin 1000 milligram (mg) and Gliclazide 30 mg fixed combination tablet in fasting state in treatment period 1 followed by single dose of Metformin 1000 mg and Gliclazide 30 mg fixed combination tablet in fed state in treatment period 2. Each treatment period was separated by a 14-day wash-out period.
  Interventions: Drug: Metformin/Gliclazide Fixed Combination
- Metformin-Gliclazide (fed), Then Metformin-Gliclazide (fasted) (Experimental): Participants received single dose of Metformin 1000 mg and Gliclazide 30 mg fixed combination tablet in fed state in treatment period 1 followed by single dose of Metformin 1000 mg and Gliclazide 30 mg fixed combination tablet in fasting state in treatment period 2. Each treatment period will be separated by a 14-day wash-out period.
  Interventions: Drug: Metformin/Gliclazide Fixed Combination

INTERVENTIONS:
Drug: Metformin/Gliclazide Fixed Combination — Participants will receive single oral dose of Metformin 1000 mg and Gliclazide 30 mg fixed combination tablet in fasting or fed state.

SUMMARY:
This study will assess the food effect on bioavailability of Metformin/Gliclazide fixed dose combination tablet in fed and fasted state.

ELIGIBILITY:
Inclusion Criteria:

* Ethnicity: Mexicans
* Weight between 55 and 95 kilogram (kg)
* Body mass index between 18 and 27 kilogram per meter square (kg/m^2)
* Nonsmokers or participants who do not smoke more than 5 cigarettes or 1 pipe a day
* Good physical and mental health based on the clinical history and physical examination
* All results from blood chemistry, hematology, and urinalysis should be within normal ranges or without clinically significant deviations as per Principal Investigator's judgment
* Hematology complete blood count [CBC]: hematocrit and hemoglobin must be above the lower limit; upper limit may range up to 15 percent (%)
* Liver Function Test range as defined in the protocol
* Electrocardiogram (12 leads) without clinically significant pathological signs
* All women of childbearing potential must have negative tests for pregnancy at screening, and at day -1 for each treatment period and at end of trial (EOT)
* Vital signs (blood pressure and pulse) in supine position within normal ranges or with clinically significant abnormalities as per the Principal Investigator's judgment
* All women of childbearing potential who are not pregnant or breastfeeding and who are using a highly effective contraceptive method for at least one month before and following dosing
* Negative result for alcohol breath test and urine test for drugs of abuse at screening and at each day -1 of the 2 treatment periods
* Negative serology tests for human immunodeficiency virus (HIV1 and HIV2 antibodies), hepatitis A (HAV), hepatitis B (HBV), hepatitis C (HCV) and venereal disease research laboratory (VDRL) test screening
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Participants who have received any investigational drug within 21 days prior to the study start
* Participants who have donated or lost 450 milliliter (mL) or more of blood within 21 days prior to the study start
* Participants with history of cardiovascular, renal, liver, metabolic, gastrointestinal, neurological, endocrine, or hematopoietic (any type of anemia) diseases; mental disease, surgery or other organic abnormalities which might affect the study of the investigational drug pharmacokinetics
* History of gastrointestinal tract surgery
* Participants with history of hypersensitivity to the study drug and/or any formulation's ingredient; history of drug induced anaphylaxis
* Participants who take any other drug 30 days before the study drug dose and for which at least seven elimination half-lives had not elapsed
* Renal failure or renal impairment assessed by using the Cockcroft-Gault formula
* Participant's disagreement or lack of capacity to communicate and cooperate with the Investigator, lack of legal capacity or limited legal capacity which prevent him/her from continuing in the study
* Refusal of the high-fat diet which is necessary to assess the food effect. Considerable deviations to the diet's normal nutritional patterns
* Participants who have smoked tobacco, having drunk alcohol, or xanthines containing beverages or food above 600 mg of caffeine a day those who have had grilled food within 24 h prior to the drug dosing
* Intake of grapefruit, orange, cranberries or their juices within 14 days prior to the drug's dosing and throughout the study
* Legal inability or limited legal capacity
* Incarcerated participants
* Participants who have been exposed to agents known as liver enzyme systems' inducers or inhibitors, or who have taken potentially toxic drugs within 30 days prior to the study
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2018-03-06 (Actual); Primary Completion 2018-04-22 (Actual); Study Completion 2018-04-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- CECYPE, Mexico City, Mexico

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period 1
Arm/Group | Metformin-Gliclazide (Fasted), Then Metformin-Gliclazide (Fed) | Metformin-Gliclazide (Fed), Then Metformin-Gliclazide (Fasted)
Started | 10 | 11
Completed | 10 | 11
Not Completed | 0 | 0
Period: Treatment Period 2
Arm/Group | Metformin-Gliclazide (Fasted), Then Metformin-Gliclazide (Fed) | Metformin-Gliclazide (Fed), Then Metformin-Gliclazide (Fasted)
Started | 10 | 11
Completed | 10 | 10
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin-Gliclazide (Fasted), Then Metformin-Gliclazide (Fed) | Metformin-Gliclazide (Fed), Then Metformin-Gliclazide (Fasted) | Total
Number analyzed (Participants) | 10 | 11 | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 37.2 (10.9) | 32.5 (8.0) | 34.7 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6
  Male | 7 | 8 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 11 | 21
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC0-inf) of Metformin and Gliclazide
Description: AUC (0-inf) is defined as the area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf).
Time Frame: Pre-dose, 0.5, 1.0, 2.0, 3.0, 4.0, 5.0, 6.0, 7.0, 8.0, 10.0, 12.0, 16.0, 24.0, 28.0, 32.0, 48.0, 72.0, 96.0, 120.0, 144.0 and 168.0 hour post-dose
Population: The Pharmacokinetics (PK) analysis set included all participants who completed the study with adequate study medication compliance, without any relevant protocol violations with respect to factors likely to affect the comparability of PK results.
Measure: Mean (Standard Deviation); unit: Nanogram*hour per milliliter (ng*h/mL)
Groups:
- Metformin-Gliclazide (Fasted): Participants received single dose of Metformin 1000 mg and Gliclazide 30 mg fixed combination tablet in fasting state in treatment period 1 or in treatment period 2.
- Metformin-Gliclazide (Fed): Participants received single dose of Metformin 1000 mg and Gliclazide 30 mg fixed combination tablet in fed state in treatment period 1 or in treatment period 2.
Arm/Group | Metformin-Gliclazide (Fasted) | Metformin-Gliclazide (Fed)
Number analyzed (Participants) | 21 | 21
Nanogram*hour per milliliter (ng*h/mL)
  Metformin | 4974.2507 (1599.3290) | 8556.7752 (2544.6658)
  Gliclazide | 21192.1682 (9220.3044) | 21815.4021 (8369.0107)
Statistical Analysis 1: Comparison: Metformin-Gliclazide (Fasted) vs Metformin-Gliclazide (Fed); Statistical Analysis for Metformin; Test type: Equivalence — Bio-equivalence Analysis was performed with Equivalence Acceptance Range for 90% Confidence Interval (CI) as 80.0% - 125.0%; Ratio of mean values = 175.6652, 90% CI 2-sided [153.7790 to 200.6664]
Statistical Analysis 2: Comparison: Metformin-Gliclazide (Fasted) vs Metformin-Gliclazide (Fed); Statistical Analysis for Gliclazide; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of mean values = 104.457, 90% CI 2-sided [97.7660 to 111.6060]

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUC0-t) of Metformin and Gliclazide
Description: AUC (0-t) is defined as the area under the plasma concentration versus time curve from time zero (pre-dose) to time of last quantifiable concentration (0-t)
Time Frame: as for outcome 1
Population: PK analysis set included all participants who completed the study with adequate study medication compliance, without any relevant protocol violations with respect to factors likely to affect the comparability of PK results.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Metformin-Gliclazide (Fasted) | Metformin-Gliclazide (Fed)
Number analyzed (Participants) | 21 | 21
ng*h/mL
  Metformin | 4722.4546 (1598.1082) | 8298.5628 (2422.9059)
  Gliclazide | 20348.8381 (9154.5509) | 20997.1704 (8244.2743)
Statistical Analysis 1: Comparison: Metformin-Gliclazide (Fasted) vs Metformin-Gliclazide (Fed); Statistical Analysis for Metformin; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of mean values = 180.7734, 90% CI 2-sided [157.0135 to 208.1287]
Statistical Analysis 2: Comparison: Metformin-Gliclazide (Fasted) vs Metformin-Gliclazide (Fed); Statistical Analysis for Gliclazide; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of mean values = 105.0818, 90% CI 2-sided [98.0047 to 112.6699]

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Metformin and Gliclazide
Description: Cmax is defined as the maximum observed plasma concentration.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Metformin-Gliclazide (Fasted) | Metformin-Gliclazide (Fed)
Number analyzed (Participants) | 21 | 21
ng/mL
  Metformin | 717.5017 (304.8105) | 870.7288 (272.6886)
  Gliclazide | 968.0305 (261.8362) | 1013.9753 (243.1601)
Statistical Analysis 1: Comparison: Metformin-Gliclazide (Fasted) vs Metformin-Gliclazide (Fed); Statistical Analysis for Metformin; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of mean values = 127.7779, 90% CI 2-sided [110.2732 to 148.0612]
Statistical Analysis 2: Comparison: Metformin-Gliclazide (Fasted) vs Metformin-Gliclazide (Fed); Statistical Analysis for Gliclazide; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of mean values = 105.4183, 90% CI 2-sided [94.5723 to 117.5081]

4. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Metformin and Gliclazide
Description: Tmax is defined as the time to reach maximum plasma concentration.
Time Frame: as for outcome 1
Population: The PK analysis set included all participants who completed the study with adequate study medication compliance, without any relevant protocol violations with respect to factors likely to affect the comparability of PK results.
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Metformin-Gliclazide (Fasted) | Metformin-Gliclazide (Fed)
Number analyzed (Participants) | 21 | 21
Hours
  Metformin | 3.6698 (0.6600) | 7.2389 (0.7693)
  Gliclazide | 6.5254 (1.7474) | 8.5238 (2.1822)

5. Secondary Outcome: Elimination Half Life (t1/2) of Metformin and Gliclazide
Description: Elimination Half Life (t1/2) is defined as the time required for the concentration or amount of drug in the body to be reduced by one-half.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Metformin-Gliclazide (Fasted) | Metformin-Gliclazide (Fed)
Number analyzed (Participants) | 21 | 21
Hours
  Metformin | 6.2547 (2.9771) | 7.4892 (8.7276)
  Gliclazide | 16.6222 (6.2627) | 17.1044 (7.5000)

6. Secondary Outcome: Apparent Volume of Distribution (Vz/f) of Metformin and Gliclazide
Description: Vz/f is defined as apparent volume of distribution during terminal phase after non-intravenous administration
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Milliliter (mL)
Arm/Group | Metformin-Gliclazide (Fasted) | Metformin-Gliclazide (Fed)
Number analyzed (Participants) | 21 | 21
Milliliter (mL)
  Metformin | 2003389.9474 (1157828.4547) | 1200933.2647 (949837.2019)
  Gliclazide | 35189.3864 (8855.9499) | 33813.7843 (6970.7706)

7. Secondary Outcome: Apparent Total Body Clearance (CL/f) of Metformin and Gliclazide From Plasma
Description: CL/f is defined as apparent total clearance of the drug from plasma after oral administration.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- Metformin-Gliclazide (Fasted): Participants received single dose of Metformin 1000 mg and Gliclazide 30 mg fixed combination tablet in fasted state in treatment period 1 or in treatment period 2.
Arm/Group | Metformin-Gliclazide (Fasted) | Metformin-Gliclazide (Fed)
Number analyzed (Participants) | 21 | 21
Liters
  Metformin | 226.79 (88.58) | 125.93 (33.92)
  Glilclazide | 1.63 (0.57) | 1.55 (0.52)

8. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Adverse event(AE) was defined as any untoward medical occurrence in participants which does not necessarily have causal relationship with treatment. AE was any unfavorable and unintended sign(including abnormal laboratory finding), symptom/disease temporally associated with use of medicinal product, whether/not considered related to medicinal product. A serious adverse event(SAE) was AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial/prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. Term TEAE is defined as AEs starting/worsening after first intake of the study drug. TEAEs included both Serious TEAEs and non-serious TEAEs.
Time Frame: Baseline up to Day 39
Population: The safety population included all participants who received at least 1 dose of the study treatment in either treatment period 1 or treatment period 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Metformin-Gliclazide (Fasted) | Metformin-Gliclazide (Fed)
Number analyzed (Participants) | 21 | 21
Participants
  Adverse Events | 8 | 7
  Serious Adverse Events (SAEs) | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Day 39
Description: The safety population included all participants who received at least 1 dose of the study treatment.
Arm/Group | Metformin-Gliclazide (Fasted) | Metformin-Gliclazide (Fed)
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 8/21 | 7/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin-Gliclazide (Fasted) (N=21) | Metformin-Gliclazide (Fed) (N=21)
Elevated triglycerides (Investigations) | 2 | 3
Elevated total bilirubin (Investigations) | 1 | 0
Elevated direct bilirubin (Investigations) | 1 | 0
Elevated indirect bilirubin (Investigations) | 1 | 0
High cholesterol (Investigations) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 3
Headache (Nervous system disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/71/NCT03467971/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/71/NCT03467971/SAP_001.pdf